CLINICAL TRIAL: NCT00285077
Title: Long-Term Safety Extension of Phase II Study EFC5286 of SR57667B in Patients With Mild-to-Moderate Alzheimer's Disease
Brief Title: Long-Term Safety Extension With SR57667B in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTS5283
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; nerve growth factors; Clinical Trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR57667B

SUMMARY:
The primary objective is to assess the long term safety/tolerability of 4 mg/day of SR57667B in comparison to placebo in patients with mild-to-moderate Alzheimer's Disease (AD).

A secondary objective is to describe the long term progression of Alzheimer's symptoms in patients treated by 4 mg/day of SR57667B.

DETAILED DESCRIPTION:
Multinational, multicenter, randomized, parallel-group, double-blind, phase II study

ELIGIBILITY:
Inclusion Criteria:

* Patients who have participated in Study EFC5286 and completed the study.
* Patient, identified caregiver and, if applicable, patient surrogate (primary relative, legal guardian, medical proxy) have given their informed written consent and are capable of following study procedures specifically for this LTS5283 extension.

Exclusion Criteria:

* Females who are pregnant or breast-feeding.
* Females of child bearing potential (premenopausal female biologically capable of becoming pregnant) must have a confirmed negative serum b-HCG pregnancy test at the screening visit,and must use an acceptable method of birth control.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2004-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Adverse events recorded quarterly.

SECONDARY OUTCOMES:
ADAS-cog, CDR, MMSE, CGIC, ADCS-ADL, NPI measured at baseline and at 2,6,9 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Serge GAUTHIER, MD, Study Chair — Scientific Advisory Committee; Jean-Marc ORGOGOZO, MD, Study Chair — Scientific Advisory Committee; Philip SCHELTENS, MD, Study Chair — Scientific Advisory Committee; Bengt WINBLAD, MD, Study Chair — Scientific Advisory Committee
Locations (7):
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Horslholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com